CLINICAL TRIAL: NCT00046735
Title: A Single-Center, Open-Label, Between-Patient, Dose-Escalation Phase 1 Study of CDC-501 In Patients With Solid Tumors
Brief Title: Phase 1 Study OF CDC-501 in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-ST-003
Record Dates: First submitted 2002-10-02; First posted 2002-10-03 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Neoplasms
Keywords: solid tumors; Revimid; CC5013; CC-5013
MeSH Terms: conditions — Neoplasms | interventions — Lenalidomide

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — The planned doses for investigation are as follows: 5, 10, and 25 mg/day. Lenalidomide will be administered as a single daily dose for 4 weeks followed by a 2-week rest period. Dosing will be in the morning at approximately the same time each day, at least 1 hour before the morning meal. Patients will be assigned to dose level in the order of study entry. No dose adjustments or suspensions are allowed during the first cycle, except discontinuation for DLT

SUMMARY:
To identify the maximum tolerated dose (MTD) and safety of CDC-501 when given in a 6-week cycle in patients with solid tumors that are refractory after standard treatment.

DETAILED DESCRIPTION:
Identify the maximum tolerated dose (MTD) and safety of CDC-501 when given in a 6-week cycle in patients with solid tumors that are refractory after standard treatment

ELIGIBILITY:
Inclusion Criteria:

1. Patient must understand and voluntarily sign an informed consent document.
2. Age 18 years at the time of signing Informed Consent
3. Histologically or cytologically documented solid tumors that are refractory to standard/conventional therapy or for which no standard/conventional therapy exists.
4. Patients must have at least one measurable or non-measurable lesion according to the RECIST Criteria (Appendix I).
5. Patient has an ECOG (Zubrod) performance status of ≤ 2.
6. Approximate life expectancy greater than 3 months.
7. Laboratory tests within these ranges:

   * Absolute neutrophil count ≥ 1,500/μlL
   * Platelet count ≥100,000/μL
   * Serum creatinine ≤1.5 mg/dL
   * Total bilirubin ≤1.5 mg/dL
   * AST (SGOT)/ALT(SGPT) ≤ 2 x upper limit of normal (ULN) or ≤ 5 x ULN if hepatic metastases present
8. The following prior treatments are allowable under this protocol:
9. Radiation, if discontinued at least 4 weeks prior to treatment under this protocol Chemotherapy, if discontinued at least 4 weeks prior to treatment under this protocol, and at least 6 weeks prior to treatment under this protocol for prior nitrosurea or mitomycin-C treatment
10. Hormonal therapy for cancer, if discontinued at least 4 weeks prior to treatment under this protocol
11. Other investigational drugs, if discontinued at least 4 weeks prior to treatment under this protocol
12. Surgery, if minor surgery occurred at least 2 weeks prior to treatment under this protocol, or at least 4 weeks since major surgery
13. Patient must be able to adhere to the study visit schedule and other protocol requirements.
14. Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test within 7 days prior to baseline. In addition, sexually active WCBP must agree to use adequate contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner).

Exclusion Criteria

1. Myocardial infarction within the previous 6 months, unstable angina,symptomatic congestive heart failure, or other significant uncontrolled cardiac arrhythmia.
2. Cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis or other significant thromboembolic event in the previous 6 months.
3. Active infection, including known human immunodeficiency virus (HIV) positivity or acquired-immunodeficiency-syndrome (AIDS)-related illness.
4. CNS metastases, unless controlled by previous radiation and the patient is neurologically stable.
5. Any serious medical condition, laboratory abnormality or psychiatric illness that would prevent the patient from signing the informed consent or limit survival to less than 3 months.
6. Pregnant or nursing females.Female patients of childbearing potential who are unwilling to use reliable contraceptive methods.
7. Any condition, including the presence of laboratory abnormalities, which in the opinion of the Investigator places the patient at unacceptable risk if he/she were to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2002-06-01 (Actual); Primary Completion 2006-08-01 (Actual); Study Completion 2006-09-28 (Actual)

PRIMARY OUTCOMES:
To identify the MTD and safety of CDC-501 when given in a 6-wk cycle of daily administration of CDC-501 for 4 wks followed by a 2-wk rest in doses of 5 mg/day up to 25 mg/day in pts with solid tumors that are refractory after standard treatment. | 6-week cycle comprising daily administration of CDC-501 for 4 weeks followed by a 2-week rest

CONTACTS AND LOCATIONS:
Overall Officials: Robert Knight, MD, Study Director — Celgene Corporation
Locations (1):
- Wake Forest University, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Miller AA, Case D, Harmon M, Savage P, Lesser G, Hurd D, Melin SA. Phase I study of lenalidomide in solid tumors. J Thorac Oncol. 2007 May;2(5):445-9. doi: 10.1097/01.JTO.0000268679.33238.67. PMID 17473661